CLINICAL TRIAL: NCT03596164
Title: An Open-Label, Extension Study of Teduglutide in Japanese Subjects With Short Bowel Syndrome Who Completed 24 Weeks of Treatment in SHP633-306 or TED-C14-004
Brief Title: An Extension Study of Teduglutide in Japanese Participants With Short Bowel Syndrome Who Completed 24 Weeks of Treatment in SHP633-306 or TED-C14-004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-307
Record Dates: First submitted 2018-06-28; First posted 2018-07-23 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; Syringes; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teduglutide 0.05 mg (Experimental): Participants will receive Teduglutide 0.05 milligram per kilogram (mg/kg) subcutaneous (SC) injection once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm until Teduglutide is commercially available, the participant's participation in this study is discontinued, or the study is discontinued.
  Interventions: Drug: Teduglutide; Device: Syringe; Device: Needle; Device: Vial Adapter for Device

INTERVENTIONS:
Drug: Teduglutide — Teduglutide 0.05 mg/kg SC injection will be administered once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm.
Device: Syringe — Teduglutide will be administered using syringe. Syringe is approved for use in Japan by PMDA.
Device: Needle — Teduglutide will be administered using needle. Needle is approved for use in Japan by PMDA.
Device: Vial Adapter for Device — Vial adapter for device is approved for use in Japan by PMDA.

SUMMARY:
The purpose of this clinical study is to evaluate the long-term safety and efficacy of teduglutide in Japanese participants with PN/IV (parenteral nutrition/intravenous)-dependent SBS (short bowel syndrome) who completed SHP633-306 or who were in the extension phase of the TED-C14-004 (NCT02340819) study.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria will be enrolled in this study:

1. Ability to voluntarily provide written, signed, and informed consent to participate in the study.
2. Completion of the SHP633-306 study or participation in TED-C14-004 (NCT02340819) Stage 3 or Stage 4.
3. Females of childbearing potential must agree to comply with the contraceptive requirements of the protocol.
4. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Japan (5):
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hyogo College of Medicine Hospital, Hyōgo
  - Tohoku University Hospital, Miyagi-Ken
  - Osaka University Hospital, Osaka
  - Yokohama Municipal Citizen's Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab470f1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Japan from 09 July 2018 to 13 January 2022.
Pre-assignment Details: Participants with a historical diagnosis with short bowel syndrome, who completed 24 weeks of treatment in core studies SHP633-306 (NCT03663582) or TED-C14-004 (NCT02340819) were enrolled and received teduglutide in this current study (SHP633-307). Total study duration were approximately 13 months for SHP633-306 (NCT03663582) and approximately 47 months for TED-C14-004 (NCT02340819).
Groups:
- SHP633-306: Teduglutide 0.05 mg/kg: Participants who completed SHP633-306 (NCT03663582) were enrolled and received teduglutide 0.05 milligram per kilogram (mg/kg), subcutaneous injection, once daily for up to approximately 30.3 months in this study.
- TED-C14-004: Teduglutide 0.05 mg/kg: Participants who were in extension phase of TED-C14-004 (NCT02340819) were enrolled and received teduglutide 0.05 mg/kg, subcutaneous injection, once daily for up to approximately 40.2 months in this study.
Period: Overall Study
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Started | 4 | 7
Completed | 3 | 6
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants in the study. Data reported in baseline measures was collected at baseline of core studies (SHP633-306 [NCT03663582] or TED-C14-004 [NCT02340819]).
Groups:
- SHP633-306: Teduglutide 0.05 mg/kg: Participants who completed SHP633-306 (NCT03663582) were enrolled and received teduglutide 0.05 mg/kg, subcutaneous injection, once daily for up to approximately 30.3 months in this study.
- Total: Total of all reporting groups
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (12.28) | 42.4 (7.21) | 41.8 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 7 | 11
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 161.10 (6.168) | 167.77 (6.735) | 165.35 (7.068)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 49.29 (10.010) | 56.01 (10.958) | 53.57 (10.660)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 18.96 (3.441) | 19.80 (3.153) | 19.49 (3.114)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Demonstrated at Least 20 Percent (%) Reduction From Baseline in Weekly Parenteral Support (PS) Volume
Description: The weekly volume was calculated as (sum of daily volumes in the diary/number of days with values)*7. Baseline data refer to the baseline of core studies (SHP633-306 [NCT03663582] or TED-C14-004 [NCT02340819]), however the time frame represents the duration for which participants were assessed in current study. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data of the Core Study.
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Number analyzed (Participants) | 4 | 7
Participants | 3 | 5

2. Primary Outcome: Change From Baseline in Weekly PS Volume
Description: as for outcome 1
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Mean (Standard Deviation); unit: liter per week (L/Week)
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Number analyzed (Participants) | 4 | 7
liter per week (L/Week) | -7.45 (7.908) | -8.67 (7.450)

3. Primary Outcome: Percent Change From Baseline in Weekly PS Volume
Description: as for outcome 1
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Number analyzed (Participants) | 4 | 7
percent change | -49.55 (41.411) | -52.52 (39.828)

4. Primary Outcome: Number of Participants Who Were Completely Weaned Off PS at End of Study (EOS)
Time Frame: From the first dose of study drug (in current study) up to EOS (up to approximately 42 months)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Number analyzed (Participants) | 4 | 7
Participants | 1 | 2

5. Primary Outcome: Change From Baseline in Days Per Week of PS
Description: Baseline data refer to the baseline of core studies (SHP633-306 [NCT03663582] or TED-C14-004 [NCT02340819]), however the time frame represents the duration for which participants were assessed in current study. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data of the Core Study.
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Number analyzed (Participants) | 4 | 7
days per week | -2.3 (3.30) | -2.0 (3.42)

6. Primary Outcome: Change From Baseline in Plasma Citrulline Levels
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Plasma samples were analyzed using a validated high-performance liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. Baseline data refer to the baseline of core studies (SHP633-306 [NCT03663582] or TED-C14-004 [NCT02340819]), however the time frame represents the duration for which participants were assessed in current study. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data of the Core Study.
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg
Number analyzed (Participants) | 4 | 7
micromoles per liter | 12.96 (5.568) | 19.15 (18.851)

7. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: From the first dose of study drug (in current study) up to EOS (up to approximately 42 months)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Total Participants: All participants who completed SHP633-306 (NCT03663582) and were in extension phase of TED-C14-004 (NCT02340819) were enrolled and received teduglutide 0.05 mg/kg, subcutaneous injection, once daily for up to approximately 40.2 months in this study.
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants
  TEAE | 4 | 7 | 11
  TESAE | 3 | 4 | 7

8. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Values
Description: as for outcome 5
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign Measurements
Description: as for outcome 5
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Description: as for outcome 5
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 0 | 0 | 0

11. Primary Outcome: Number of Participants Who Reported Positive Specific Antibodies to Teduglutide at EOS
Time Frame: From the first dose of study drug (in current study) up to EOS (up to approximately 42 months)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 3 | 4 | 7

12. Primary Outcome: Change From Baseline in 48-Hour Urine Output
Description: as for outcome 5
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Mean (Standard Deviation); unit: Milliliter per day (mL/day)
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Milliliter per day (mL/day) | 428.8 (286.57) | 308.6 (589.36) | 352.3 (486.54)

13. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Body Weight Measurements
Description: as for outcome 5
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in BMI
Description: as for outcome 5
Time Frame: Baseline (core study) up to approximately 40.2 months (duration of assessment in the current study)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Clinically Significant Colonoscopy/Sigmoidoscopy Results
Time Frame: From the first dose of study drug (in current study) up to EOS (up to approximately 42 months)
Population: The safety population included all enrolled participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
Number analyzed (Participants) | 4 | 7 | 11
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were defined as AEs that started on or after the first dose of study drug (in current study) up to approximately 42 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | SHP633-306: Teduglutide 0.05 mg/kg | TED-C14-004: Teduglutide 0.05 mg/kg | Total Participants
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/7 | 1/11
Serious Adverse Events (participants affected / at risk) | 3/4 | 4/7 | 7/11
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SHP633-306: Teduglutide 0.05 mg/kg (N=4) | TED-C14-004: Teduglutide 0.05 mg/kg (N=7) | Total Participants (N=11)
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Device breakage (Product Issues) | 1 | 0 | 1
Device occlusion (Product Issues) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 4 | 4
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Subclavian vein occlusion (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SHP633-306: Teduglutide 0.05 mg/kg (N=4) | TED-C14-004: Teduglutide 0.05 mg/kg (N=7) | Total Participants (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 2
Anal erosion (Gastrointestinal disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
C-reactive protein increased (Investigations) | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Device related infection (Infections and infestations) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Dry eye (Eye disorders) | 0 | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 5
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Selenium deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Vaccination site pain (General disorders) | 1 | 1 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03596164/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT03596164/SAP_002.pdf